CLINICAL TRIAL: NCT02421900
Title: Analysis of the Role of T-cell Response in Patients With Atrial Fibrillation for Clinical Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0090
Record Dates: First submitted 2015-04-08; First posted 2015-04-21 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 40cc blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- group 1: Atrial fibrillation patients
  Interventions: Other: radio-frequency catheter ablation of atrial fibrillation

INTERVENTIONS:
Other: radio-frequency catheter ablation of atrial fibrillation — radio-frequency catheter ablation of atrial fibrillation

SUMMARY:
The purpose of this study is 1) to characterize T-cell response in patients with atrial fibrillation, and 2) to analyze the changes of T-cell response after radio-frequency catheter ablation of atrial fibrillation. First, immune-phenotyping and cytokine profiling of T cells from patients with atrial fibrillation will performed. Next the difference of T-cell immunity among various type of atrial fibrillation patients will be analyzed. Finally the changes of T-cell response and cytokines after radio-frequency catheter ablation of atrial fibrillation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who consent with study
* patients with age more than19
* patients who undergoing catheter ablation of atrial fibrillation due to symptomatic, drug refractory atrial fibrillation

Exclusion Criteria:

* Patients who do not agree with study inclusion
* Permanent AF refractory to electrical cardioversion
* AF with rheumatic valvular disease
* Patients with left atrial diameter greater than 60mm
* Patients with age less than 19
* Patient with malignant tumor and chronic infection disease
* Patient are given immune inhibitor and steroidal anti-inflammatory drug within 2weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The frequency (%) of specific marker-expressing cells among CD4 or CD8 T-subsets | 1 year
  * Immunosenescence marker: CD28, CD57
  * Activation marker: CD38, HLA-DR
  * Differentiation marker: CCR7, CD45RA

SECONDARY OUTCOMES:
The frequency (%) of cytokine-secreting cells among CD4 or CD8 T-subsets | 1 year
  * Proinflammatory cytokine: IFN-gamma, TNF-alpha
  * Cytotoxic molecule: granzyme B, perforin

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea